CLINICAL TRIAL: NCT00755313
Title: Effects of Chemotherapy on Brain Structure and Function
Brief Title: Effects of Chemotherapy on the Brain in Women With Newly Diagnosed Early-Stage Breast Cancer
Status: Completed | Type: Observational
Sponsor: University of California, San Francisco (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: CDR0000613050; UCSF-06803; UCSF-H6961-29940-02B
Record Dates: First submitted 2008-09-17; First posted 2008-09-18 (Estimated); Last update posted 2017-11-24 (Actual); Status verified 2017-11

CONDITIONS: Breast Cancer; Chemotherapeutic Agent Toxicity; Cognitive/Functional Effects; Fatigue; Long-term Effects Secondary to Cancer Therapy in Adults; Neurotoxicity; Psychosocial Effects of Cancer and Its Treatment
Keywords: cognitive/functional effects; fatigue; long-term effects secondary to cancer therapy in adults; psychosocial effects of cancer and its treatment; chemotherapeutic agent toxicity; neurotoxicity; stage IA breast cancer; stage IB breast cancer; stage II breast cancer; stage IIIA breast cancer; stage IIIB breast cancer; stage IIIC breast cancer; estrogen receptor-negative breast cancer; estrogen receptor-positive breast cancer; progesterone receptor-negative breast cancer; progesterone receptor-positive breast cancer
MeSH Terms: conditions — Breast Neoplasms; Fatigue; Neurotoxicity Syndromes | interventions — Trastuzumab; Aromatase Inhibitors; Carboplatin; Cyclophosphamide; Docetaxel; Doxorubicin; Mental Status and Dementia Tests; Magnetic Resonance Spectroscopy; Fluorodeoxyglucose F18

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Biological: trastuzumab
Drug: aromatase inhibition therapy
Drug: carboplatin
Drug: cyclophosphamide
Drug: docetaxel
Drug: doxorubicin hydrochloride
Other: metabolic assessment
Other: questionnaire administration
Other: study of socioeconomic and demographic variables
Procedure: cognitive assessment
Procedure: positron emission tomography
Radiation: fludeoxyglucose F 18

SUMMARY:
RATIONALE: Gathering information over time from laboratory tests, imaging scans, and assessment tests may help doctors learn more about the side effects of chemotherapy and plan the best treatment.

PURPOSE: This clinical trial is studying the effects of chemotherapy on the brain in women with newly diagnosed early-stage breast cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To prospectively evaluate the acute (1 month after chemotherapy) and relatively long-term (18 months after chemotherapy) effects of standard-dose chemotherapy and/or hormonal therapy with aromatase inhibition on brain function using positron emission tomography (PET) and the glucose metabolism tracer fludeoxyglucose F 18 in women with newly diagnosed, early stage breast cancer.

Secondary

* To evaluate the acute and relatively long-term effects of chemotherapy and/or hormonal therapy on MRI measurements of hippocampal volume, cortical grey matter volume, white matter signal hyperintensities, ventricular volume, and whole brain volume in these patients.
* To evaluate the acute and relatively long-term effects of chemotherapy and/or hormonal therapy with aromatase inhibition on cognitive function in these patients.
* To explore the characteristics of these patients that renders them more vulnerable to chemotherapy and/or estrogen suppression-induced cognitive decline.

OUTLINE: Patients are stratified according to planned adjuvant chemotherapy (chemotherapy and hormonal therapy vs hormonal therapy vs chemotherapy vs no therapy) and the hormone receptor status (positive vs negative).

Patients (groups A-C) undergo bioavailable estradiol measurements, PET scans, and MRI scans at baseline and 1 and 18 months after treatment. Patients also undergo cognitive, neuropsychological, sociodemographic, and quality of life assessments using a battery of study tests and questionnaires at baseline and at 1, 9, and 18 months after treatment. Group D participants (controls) undergo the same testing at equivalent intervals.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of breast cancer, meeting 1 of the following criteria:

  * Group A

    * Stage I, II, or III invasive disease
    * Hormone receptor-positive disease
    * Planned adjuvant chemotherapy including an anthracycline and taxane using either dose-dense or docetaxel, doxorubicin hydrochloride, and cyclophosphamide (TAC) regimens with or without trastuzumab (Herceptin®) for 4 months; docetaxel and cyclophosphamide (TC) with or without trastuzumab for 3 months; doxorubicin hydrochloride and cyclophosphamide (AC) for 3 months; or doxorubicin hydrochloride, carboplatin, and trastuzumab (TCH) for 4 months (trastuzumab may be given for 1 year and is not considered chemotherapy for the purpose of this study)
    * Planned treatment with adjuvant aromatase inhibitors (AI) for 5 years
  * Group B

    * Stage I or II invasive disease
    * Planned treatment with adjuvant AI with or without radiotherapy
  * Group C

    * Stage I, II, or III disease
    * Hormone-receptor negative
    * Planned adjuvant chemotherapy as in group A
    * No treatment with AI planned
  * Group D

    * Healthy controls free of any major medical or psychiatric disorders
    * Not taking prescription medications, including hormone-replacement therapy, or other substances that might influence performance on neuropsychological tests
    * Balanced with the patient groups on age, education, ethnicity, and sociodemographic background

PATIENT CHARACTERISTICS:

* No history of psychiatric illness other than minor depression
* No history of psychiatric illness other than minor depression in immediate family members
* No history of neurologic disease
* No history of drug or alcohol abuse
* No significant medical illness other than breast cancer
* No heart pacemaker or metallic implants or particles in the body
* No heart rhythm disturbance
* No claustrophobia
* No prior serious head injury
* No tattoos or permanent cosmetics
* No unremovable body jewelry
* No cognitive impairment
* Able to read and speak English
* No condition that compromises compliance with the objectives and procedures of this study, as judged by the principal investigator

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* No prior chemotherapy, CNS radiotherapy, or intrathecal therapy
* Premenopausal women receiving aromatase inhibitors must also be receiving ovarian suppression
* No concurrent narcotics or major antipsychotic medications that may impair cognition

Ages: 35 Years to 80 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: women with newly diagnosed, early stage breast cancer
Sampling Method: Probability Sample
Enrollment: 81 (Actual)
Dates: Start 2007-05; Primary Completion 2012-09 (Actual); Study Completion 2014-06-06 (Actual)

PRIMARY OUTCOMES:
Change in glucose metabolism | Up to 18 months after treatment

SECONDARY OUTCOMES:
MRI measures of the brain (hippocampal volume, cortical gray matter volume, white matter signal hyperintensities, ventricular volume, whole brain volume) | Up to 18 months after treatment
Measures of cognitive function over time by Wechsler memory scale, word list memory, Stroop Color Word Test, Boston Naming Test, verbal fluency, FACIT-B functional assessment, Mini Mental State Exam, Hamilton Depression Rating Scale (Ham-D), Beck De ... | Up to 18 months after treatment
Cognitive assessments over time by FACIT-B, Ham-D, BDI-II, STAI, FSI, and MASQ, demographic and medical data | Up to 18 months after treatment

CONTACTS AND LOCATIONS:
Overall Officials: Hope S. Rugo, MD, Principal Investigator — University of California, San Francisco
Locations (1):
- UCSF Helen Diller Family Comprehensive Cancer Center, San Francisco, California, United States